CLINICAL TRIAL: NCT05539495
Title: Exercise Recovery From Persistent Major Depression in a UK Tertiary Care Centre: A Qualitative Thematic Analysis of Barriers and Drivers to Participation in a Structured Group Exercise Program
Brief Title: Exercise Recovery From Persistent Depression: A Thematic Analysis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Nottingham (Other)
Collaborators: Nottinghamshire Healthcare NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 22032
Record Dates: First submitted 2022-09-05; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Major Depressive Disorder; Depression Moderate; Depression Severe
Keywords: Exercise; Barriers; Facilitators
MeSH Terms: conditions — Depressive Disorder, Major; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Depression is a leading cause of disability worldwide and poses a large economic burden in the UK. There is evidence that exercise is beneficial in the management of depression and NICE now recommends group exercise programs as a treatment for people with mild and moderate-severe depression. Research shows that patients with severe depression are less likely to engage in exercise than patients with mild to moderate depression. There is little evidence, however, on the barriers and drivers to participation in such programs experienced by patients with depression; leading to uncertainty in the most effective way to implement these programs. We aim to analyse accounts of patients who have been referred to or participated in the Exercise Recovery Group (ERG), a group exercise program at the Nottingham Specialist Depression Service (NSDS). The NSDS is a tertiary unit where referred patients have suffered moderate-severe, persistent clinical depression. Eligible participants will be patients with persistent major depression who have agreed to referral to the ERG at the NSDS and who are able to provide informed consent. Participants will undergo a one-off 60 minute meeting via MS Teams, including an in-depth semi-structured interview on their experience as well as self-completion questionnaires assessing demographics, depression, anxiety and shame. Transcripts of the interviews will be subject to qualitative thematic analysis addressing questions on barriers and drivers of exercise treatment in depression; and the perceived impact of an exercise group on the individual participating. Themes will be developed to give an account of these questions, supported by anonymised quotes from the transcripts. The questionnaire data (on demographics, depression, anxiety, shame) will be used to characterise the group, in order to help assess directness of the evidence provided for other clinical populations; ultimately helping clinicians to implement exercise groups for depression that are acceptable for patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent major depression
* Patients who have at least agreed to referral to the Exercise Recovery Group within the previous 24 months
* Patients who are able to provide informed consent.

Exclusion Criteria:

* Patients with a main diagnosis of Bipolar Disorder.
* Patients who cannot speak fluently in English.
* Patients without an email account or access to an electronic device that could be used for the MS Teams meeting.
* Patients who are younger than 18-years-old. There is no upper age limit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with persistent major depression who have at least agreed to referral to the Exercise Recovery Group at the Nottingham Specialist Depression Service within the previous 24 months
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
What are the barriers and drivers to using exercise as a treatment for persistent major depression? via thematic analysis of semi-structured interview. | 12 months
  Semi-structured interview transcripts will be subject to a qualitative thematic analysis with simple descriptive statistics (via demographic questionnaire, PHQ9, GAD7, and ESS) to characterise the sample and support any anonymised quotes. Analysis of interviews will use a standard Qualitative software package (NVivo version 12) to conduct thematic analysis through an iterative process of coding, organising coding into themes, reviewing themes, and generating a final thematic narrative with reference to the research question. We will use both deductive and inductive elements in the thematic analysis.

SECONDARY OUTCOMES:
How do these barriers and drivers operate at different stages of 'participation', including contemplation of group participation; and within group participation? via thematic analysis of semi-structured interview. | 12 months
  Semi-structured interview transcripts will be subject to a qualitative thematic analysis with simple descriptive statistics (via demographic questionnaire, PHQ9, GAD7, and ESS) to characterise the sample and support any anonymised quotes. Analysis of interviews will use a standard Qualitative software package (NVivo version 12) to conduct thematic analysis through an iterative process of coding, organising coding into themes, reviewing themes, and generating a final thematic narrative with reference to the research question. We will use both deductive and inductive elements in the thematic analysis.
What is the perceived impact of an exercise group on the individual participating, including positive and negative effects? via thematic analysis of semi-structured interview. | 12 months
  Semi-structured interview transcripts will be subject to a qualitative thematic analysis with simple descriptive statistics (via demographic questionnaire, PHQ9, GAD7, and ESS) to characterise the sample and support any anonymised quotes. Analysis of interviews will use a standard Qualitative software package (NVivo version 12) to conduct thematic analysis through an iterative process of coding, organising coding into themes, reviewing themes, and generating a final thematic narrative with reference to the research question. We will use both deductive and inductive elements in the thematic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Nixon, BSc,MMedSci,MBBS,DM,FRCPsych, Principal Investigator — University of Nottingham
Locations (1):
- Nottinghamshire Healthcare NHS Foundation Trust, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Background] Braun V, Clarke V. To saturate or not to saturate? Questioning data saturation as a useful concept for thematic analysis and sample-size rationales. https://doi.org/101080/2159676X20191704846 [Internet]. 2019 [cited 2022 Apr 28];13(2):201-16.
- [Background] Depression [Internet]. [cited 2022 Apr 17].
- [Background] Al-Harbi KS. Treatment-resistant depression: therapeutic trends, challenges, and future directions. Patient Prefer Adherence. 2012;6:369-88. doi: 10.2147/PPA.S29716. Epub 2012 May 1. PMID 22654508
- [Background] Coronavirus and depression in adults, Great Britain - Office for National Statistics [Internet]. [cited 2022 Apr 17].
- [Background] Mcdaid D, Park A-L, Davidson G, John A, Knifton L, Morton A, et al. Mental Health Foundation Shari McDaid, Mental Health Foundation, Mental Health Foundation Naomi Wilson. Ment Heal Found. 2022;
- [Background] Knapen J, Vancampfort D, Morien Y, Marchal Y. Exercise therapy improves both mental and physical health in patients with major depression. Disabil Rehabil. 2015;37(16):1490-5. doi: 10.3109/09638288.2014.972579. Epub 2014 Oct 24. PMID 25342564
- [Background] Doose M, Ziegenbein M, Hoos O, Reim D, Stengert W, Hoffer N, Vogel C, Ziert Y, Sieberer M. Self-selected intensity exercise in the treatment of major depression: A pragmatic RCT. Int J Psychiatry Clin Pract. 2015;19(4):266-75. doi: 10.3109/13651501.2015.1082599. Epub 2015 Sep 23. PMID 26265421
- [Background] Schuch FB, Vasconcelos-Moreno MP, Borowsky C, Zimmermann AB, Rocha NS, Fleck MP. Exercise and severe major depression: effect on symptom severity and quality of life at discharge in an inpatient cohort. J Psychiatr Res. 2015 Feb;61:25-32. doi: 10.1016/j.jpsychires.2014.11.005. Epub 2014 Nov 21. PMID 25439084
- [Background] Schuch FB, Stubbs B. The Role of Exercise in Preventing and Treating Depression. Curr Sports Med Rep. 2019 Aug;18(8):299-304. doi: 10.1249/JSR.0000000000000620. PMID 31389872
- [Background] Schuch FB, Vancampfort D, Rosenbaum S, Richards J, Ward PB, Stubbs B. Exercise improves physical and psychological quality of life in people with depression: A meta-analysis including the evaluation of control group response. Psychiatry Res. 2016 Jul 30;241:47-54. doi: 10.1016/j.psychres.2016.04.054. Epub 2016 Apr 26. PMID 27155287
- [Background] Xie Y, Wu Z, Sun L, Zhou L, Wang G, Xiao L, Wang H. The Effects and Mechanisms of Exercise on the Treatment of Depression. Front Psychiatry. 2021 Nov 5;12:705559. doi: 10.3389/fpsyt.2021.705559. eCollection 2021. PMID 34803752
- [Background] NATIONAL INSTITUTE FOR HEALTH AND CARE EXCELLENCE Guideline Depression in adults Draft for consultation, November 2021 [Internet]. [cited 2022 May 9]. Available from: https://www.nice.org.uk/guidance/GID-
- [Background] Monteiro FC, Schuch FB, Deslandes AC, Mosqueiro BP, Caldieraro MA, Fleck MPA. Factors associated with adherence to sports and exercise among outpatients with major depressive disorder. Trends Psychiatry Psychother. 2021 Apr-Jun;43(2):108-115. doi: 10.47626/2237-6089-2019-0109. Epub 2021 Jun 15. PMID 34139115
- [Background] Stanton R, Reaburn P. Exercise and the treatment of depression: a review of the exercise program variables. J Sci Med Sport. 2014 Mar;17(2):177-82. doi: 10.1016/j.jsams.2013.03.010. Epub 2013 Apr 18. PMID 23602562
- [Background] Morriss R, Garland A, Nixon N, Guo B, James M, Kaylor-Hughes C, Moore R, Ramana R, Sampson C, Sweeney T, Dalgleish T; NIHR CLAHRC Specialist Mood Disorder Study Group. Efficacy and cost-effectiveness of a specialist depression service versus usual specialist mental health care to manage persistent depression: a randomised controlled trial. Lancet Psychiatry. 2016 Sep;3(9):821-31. doi: 10.1016/S2215-0366(16)30143-2. Epub 2016 Aug 3. PMID 27498098
- [Background] Online surveys [Internet]. [cited 2022 May 9]. Available from: https://www.onlinesurveys.ac.uk/
- [Background] HRA N. Seeking Consent in COVID-19 Research. 2020.
- [Background] PHQ-9 Depression Test Questionnaire | Patient [Internet]. [cited 2022 May 9]. Available from: https://patient.info/doctor/patient-health-questionnaire-phq-9
- [Background] GAD7 Anxiety Test Questionnaire | Patient [Internet]. [cited 2022 May 9]. Available from: https://patient.info/doctor/generalised-anxiety-disorder-assessment-gad-7
- [Background] Andrews B, Qian M, Valentine JD. Predicting depressive symptoms with a new measure of shame: The Experience of Shame Scale. Br J Clin Psychol. 2002 Mar;41(Pt 1):29-42. doi: 10.1348/014466502163778. PMID 11931676
- [Background] Braun V, Clarke V. Using thematic analysis in psychology. Qual Res Psychol. 2006 Jan;3(2):77-101.